CLINICAL TRIAL: NCT02194296
Title: An Open Label, Randomised, Two-way Crossover Study in Healthy Female and Male Volunteers to Evaluate the Relative Bioavailability of a 20 mg Ambroxol Hydrochloride Lozenge in Comparison to 30 mg Ambroxol Hydrochloride Syrup (Mucosolvan®)
Brief Title: Relative Bioavailability of Ambroxol Hydrochloride Lozenge in Comparison to Ambroxol Hydrochloride Syrup (Mucosolvan®) in Healthy Female and Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18.479
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- Ambroxol hydrochloride - lozenge (Experimental)
  Interventions: Drug: Ambroxol hydrochloride - lozenge
- Ambroxol hydrochloride - syrup (Active Comparator): Mucosolvan®
  Interventions: Drug: Ambroxol hydrochloride - syrup

INTERVENTIONS:
Drug: Ambroxol hydrochloride - lozenge
  Arms: Ambroxol hydrochloride - lozenge
Drug: Ambroxol hydrochloride - syrup
  Arms: Ambroxol hydrochloride - syrup

SUMMARY:
Study to investigate the relative bioavailability of a 20 mg ambroxol hydrochloride lozenge compared to 30 mg ambroxol hydrochloride syrup (Mucosolvan®) after dose normalisation

ELIGIBILITY:
Inclusion Criteria:

* All participants in the study should be healthy males and females
* Ages range from 18 to 55 years
* Broca Index of > -20% and < +20 %
* Prior to admission of study all volunteers will have given their written informed consent in accordance with Good Clinical Practice (GCP) and the local legislation
* Each subject will have his medical history taken and will receive a complete medical examination (incl. blood pressure and pulse rate measurements) as well as a 12-lead Electrocardiogram (ECG)
* Haematopoietic, hepatic and renal function tests will be carried out in the laboratory
* The subjects will fast for 12 hours before collection of specimens for all laboratory evaluations. The above mentioned examinations will be performed within 14 days before the first administration to the test substance

Exclusion Criteria:

* Volunteers will be excluded from the study if the results of the medical examination or laboratory test are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic immunological or hormonal disorders
* Volunteers with diseases of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Volunteers who have taken a drug with a long half-life (>= 24 hours) within one month before enrolment in the study
* Volunteers who received any other drugs which might influence the results of the trial during the week previous to the start of the study
* Volunteers who have participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who smoke (more than 10 cigarettes or 3 cigars or 3 pipes/day)
* Volunteers who are not able to refrain from smoking on study days
* Volunteers who drink more than 60 g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who have participated in excessive physical activities (e.g. competitive sports) within the last week before the study
* Volunteers who have donated blood (> 100 ml) within the last 4 weeks prior to administration

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. sterilization, Intrauterine Devices (IUD), oral contraceptives
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 1999-06; Primary Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed concentration of the analyte in plasma) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose

SECONDARY OUTCOMES:
Tmax (Time from dosing to the maximum concentration of the analyte in plasma) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
AUC0-t (Total area under the plasma concentration-time curve from time of administration to the last quantifiable drug concentration) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
λz (Terminal rate constant in Plasma) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
t½ (Terminal half-life of the analyte in plasma) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
MRTtot (Total mean residence time ) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | predose, 0.25, 0.5,.0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 36 hours postdose
Number of patients with adverse events | up to 26 days
Number of patients with clinically significant changes in vital signs | up to 26 days
Number of patients with abnormal changes in laboratory parameters | up to 26 days